CLINICAL TRIAL: NCT05465889
Title: Comparison of the Efficacy and Safety of Oral Sulfate Solution and 3-liter Polyethylene Glycol on Bowel Preparation Before Colonoscopy: a Multicenter Randomized Controlled Phase III Trial
Brief Title: Efficacy and Safety of Oral Sulfate Solution on Bowel Preparation for Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Hospital of Integrated Traditional Chinese and Western Medicine (Unknown); China-japan Friendship Hospital, Jilin University (Unknown); Beijing Hospital (Other Government); The First Affiliated Hospital of Nanchang University (Other); Zhongshan Hospital Xiamen University (Other); Henan Provincial People's Hospital (Other); Hebei Provincial People's Hospital (Unknown); Shandong University Qilu Hospital (Unknown)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: SPMS oral solution
Record Dates: First submitted 2022-02-21; First posted 2022-07-20 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Bowel Preparation for Colonoscopy
Keywords: colonoscopy; Bowel preparation; Sodium Potassium and Magnesium Sulfate; polyethylene glycol
MeSH Terms: interventions — glycoprep

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OSS group (Experimental): Bowel preparation for colonoscopy was performed using oral sulfate solution as laxative
  Interventions: Drug: Oral sulfate solution (OSS)
- Polyethylene glycol group (Active Comparator): Bowel preparation for colonoscopy was performed using polyethylene glycol as laxative
  Interventions: Drug: Polyethylene Glycol Electrolyte

INTERVENTIONS:
Drug: Oral sulfate solution (OSS) — OSS contained 17.5 g sodium sulfate, 3.13 g potassium sulfate, 1.6 g magnesium sulfate, and flavoring agents in an aqueous liquid form supplied in a 177 mL bottle. Take 177ml sodium, potassium and magnesium sulfates oral solution (diluted to 480ml) within 30 minutes 14-16 hours before colonoscopy, followed by two doses of 480ml warm water within 1 hour; Repeat the procedure 3-4 hours before colonoscopy.
  Arms: OSS group
Drug: Polyethylene Glycol Electrolyte — Take 1000 ml polyethylene glycol electrolyte solution within 1 hour at 8 p.m. the day before colonoscopy; take 2000 ml polyethylene glycol electrolyte solution within 2 hour 4-6 hours before colonoscopy.
  Arms: Polyethylene glycol group

SUMMARY:
To evaluate whether oral sulfate solution used for colon cleaning in adults prior to colonoscopy was not inferior to 3-liter polyethylene glycol in the proportion of subjects with BBPS score (total colon) ≥6 after colonoscopy

DETAILED DESCRIPTION:
Polyethylene glycol (PEG) is the most widely used laxative at present, but volume of oral PEG liquid is large and the taste of PEG is not good, so some patients could not take enough laxative to complete bowel preparation. Oral sulfate solution containing sodium sulfate, magnesium sulfate, and potassium sulfate as active ingredients was developed as osmotic laxative for bowel cleansing preparation. The OSS works on the principle that sulfate is a poorly absorbed anion. Compared to traditional magnesium sulfate solution, OSS not only tastes better, but also reduces the occurrence of electrolyte disturbances.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate and sign informed consent;
* Scheduling screening, surveillance, and diagnostic colonoscopy;
* Necessary body fluid and blood electrolyte balance (the test values of potassium, sodium, chlorine, calcium and magnesium in blood biochemistry during screening period should not exceed 10% of the normal range).

Exclusion Criteria:

* Subjects who used drugs that affect gastrointestinal dynamics, affect kidney function, or increase the risk of fluid retention or electrolyte disorders within 7 days before the start of the trial;
* Subjects with serious cardiac and cerebrovascular diseases, bronchial and lung diseases, suffering from metabolic disease or endocrine disease, abnormal blood clotting mechanism, malignant tumor, electrolyte abnormalities, epilepsy, Renal or liver dysfunction;
* Subjects with confirmed or suspected gastrointestinal obstruction, gastric retention, gastroparesis, gastric emptying disorder or acute gastrointestinal bleeding;
* Subjects with acute severe colitis (such as active severe inflammatory bowel disease, acute bacterial dysentery, diverticulitis, etc.);
* Subjects with a history of major gastrointestinal surgery (e.g. gastric bypass, gastric septal surgery, colostomy, colectomy, etc.);
* Subjects with constipation or suspected severe gastric motility disorder;
* Women with positive pregnancy tests or pregnancy plans, and women in lactation;
* Subjects who have participated in any other clinical trials within the last 3 months;
* Subjects with any other conditions that the investigator considered inappropriate for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Bowel preparation adequate rate | 30 minutes
  Proportion of subjects with total Boston bowel preparation scale (BBPS) score (total colon) ≥6.

SECONDARY OUTCOMES:
Boston bowel preparation scale (BBPS) score | 30 minutes
  The BBPS scoring rules: 0, unprepared colon segment with mucosa not seen because of solid stool that cannot be cleared; 1, portion of mucosa of the colon segment seen, but other areas of the colon segment are not well seen because of staining, residual stool, and/or opaque liquid; 2, minor amount of residual staining, small fragments of stool, and/or opaque liquid, but mucosa of colon segment is seen well; 3, entire mucosa of colon segment seen well, with no residual staining, small fragments of stool, or opaque liquid. the higher the score, the better the quality of bowel preparation.
  3 intestinal segments were scored separately: the right side of the colon (including the cecum and ascending colon), the transverse section of the colon (including the hepatic and splenic flexures), and the left side of the colon (including the descending colon, sigmoid colon, and rectum).
  Total BBPS score (0-9, the higher the score, the better the quality of bowel preparation).
Acceptability of laxatives by questionnaire survey | 12 hours
  The proportion of people who accept the laxative. Level I: the laxative has good taste and is easy to take; the intestinal clearing fluid is drunk smoothly; the intestinal preparation process is easily tolerated; Level II: The laxative has a general taste and is easy to take. The intestinal fluid is basically drunk on time, and the intestinal preparation process is barely tolerated; Level III: unacceptable laxative taste, difficult to take medicine, unable to drink the clear bowel fluid on time, intolerable bowel preparation process, refuse similar experience in the future. Under level I and Level II, the laxative was considered to be acceptable. Under level III, the laxative was considered not to be acceptable.
Colonoscopy completion rate | 30 minutes
  Proportion of subjects receiving complete colonoscopy
Incidence of laxative-related adverse events assessed by clinical examinations | 8 days
  Physical examination (skin, mucous membranes, lymph nodes, head, neck, chest, abdomen, limbs), vital signs (temperature, respirations, heart rate, blood pressure), blood routine, urine routine, blood biochemistry (DBIL, TBIL, UREA, Cr, AST, ALT, TP, ALB, GLU, TG, TC, CK, ALP, K, Na, Cl, Ca, Mg, UA), coagulation function, and 12-lead electrocardiogram were performed within 7 days before taking laxatives. The clinical examinations were repeated on the same day after the colonoscopy. All abnormal changes in clinical examination results will be assessed by clinical specialists to determine if they are related to laxative intake. Incidence was calculated as the number of subjects with laxative-related adverse events divided by the total number of subjects.

CONTACTS AND LOCATIONS:
Overall Officials: li.zhaoshen@hotmail.com li.zhaoshen@hotmail.com, M.D., Principal Investigator — Changhai Hospital, Naval Medical University
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kluge MA, Williams JL, Wu CK, Jacobson BC, Schroy PC 3rd, Lieberman DA, Calderwood AH. Inadequate Boston Bowel Preparation Scale scores predict the risk of missed neoplasia on the next colonoscopy. Gastrointest Endosc. 2018 Mar;87(3):744-751. doi: 10.1016/j.gie.2017.06.012. Epub 2017 Jun 23. PMID 28648575
- [Background] Johnson DA, Barkun AN, Cohen LB, Dominitz JA, Kaltenbach T, Martel M, Robertson DJ, Boland CR, Giardello FM, Lieberman DA, Levin TR, Rex DK; US Multi-Society Task Force on Colorectal Cancer. Optimizing adequacy of bowel cleansing for colonoscopy: recommendations from the US multi-society task force on colorectal cancer. Gastroenterology. 2014 Oct;147(4):903-24. doi: 10.1053/j.gastro.2014.07.002. No abstract available. PMID 25239068
- [Derived] Pan P, Zhao S, Wang S, Song Y, Gu L, Chen Y, Zhao J, Lu L, Li X, Xu H, Liu G, Li Y, Xu L, Wang J, Li Z, Bai Y. Comparison of the efficacy and safety of an oral sulfate solution and 3-L polyethylene glycol on bowel preparation before colonoscopy: a phase III multicenter randomized controlled trial. Gastrointest Endosc. 2023 Dec;98(6):977-986.e14. doi: 10.1016/j.gie.2023.06.070. Epub 2023 Jul 6. PMID 37422241